CLINICAL TRIAL: NCT03090243
Title: The Effects of Virtual Colonoscopy on Intraocular Pressure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shlomo gavrielli (Other)
Responsible Party: Sponsor-Investigator, Shlomo gavrielli, Doctor of medicine, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Other Study IDs: 0543-16-RMC
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Intraocular Pressure Disorder
Keywords: Glaucoma; Intraocular pressure; Colonoscopy; Virtual Colonoscopy; Valsalva
MeSH Terms: conditions — Glaucoma | interventions — Colonography, Computed Tomographic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Group: measurements of IOP before and after virtual colonoscopy
  Interventions: Device: Virtual colonoscopy

INTERVENTIONS:
Device: Virtual colonoscopy — Inserting a Foley catheter through the anus, and gas inflating of the bowel.

SUMMARY:
Our trial examined the intraocular pressure measurements differences, before and after virtual colonoscopy examination.

DETAILED DESCRIPTION:
Glaucoma is a complicated disease in which damage to the optic nerve leads to progressive, irreversible vision loss. Glaucoma is the second leading cause of blindness and associated with elevated intraocular pressure (IOP) as a major risk factor.

IOP is influenced by many factors, including ethnicity, heredity, various chemical substances (existing body and external body like drugs), physical changes (postures, neural and vascular autoregulation) and more.

Virtual colonoscopy is a common screening test for the early detection and diagnosis of colon cancer. The test is performed by computed tomography (CT) after inflating the colon with carbon dioxide (CO2) gas. The procedure is performed by inserting a Foley catheter through the anus. As a result of gas inflating of the bowel, consequently, there is an increase in the abdominal pressure.

Raising intra-abdominal pressure may cause a rise in intraocular pressure. The aim of this research is to examine the changes in IOP before and after the virtual colonoscopy, with the aim to improve the understanding of the relationship between intra-abdominal pressure and IOP.

The study will include 100 patients, men and women, that are scheduled for virtual colonoscopy test both in a hospital and in ambulatory.

ELIGIBILITY:
Inclusion Criteria:

* Participants: men and women.
* Age ≥ 18 years.
* directed by a gastroenterologist to examine colonoscopy for diagnosing colon pathology (either screening, follow-up routine or after surgery).
* patients who want to participate which are able to understand and sign, an informed consent to participate in research.

Exclusion Criteria:

* Exclusion recruitment criteria:
* Family History of Glaucoma first-degree relatives.
* patients suffering from known eye diseases, except for refractive disorders, strabismus or amblyopia, and do not take any eye care on a regular basis.
* patients with a known allergy for Localin drops.
* patients who do not want to participate or are unable to understand or sign an informed consent to participate in research.

Exclusion criteria from the study:

* The researcher doctor may remove a participant from the study if he impressed, of strong health impairments resulting from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the study include:
  Participants: men and women. Age ≥ 18 years. directed by a gastroenterologist to examine colonoscopy for diagnosing colon pathology (either screening, follow-up routine or after surgery).
  patients who want to participate which are able to understand and sign, an informed consent to participate in research.
  Exclusion recruitment criteria:
  Family History of Glaucoma first-degree relatives. patients suffering from known eye diseases, except for refractive disorders, strabismus or amblyopia, and do not take any eye care on a regular basis.
  patients with a known allergy for Localin drops. patients who do not want to participate or are unable to understand or sign an informed consent to participate in research.
  Exclusion criteria from the study: The researcher doctor may remove a participant from the study if he impressed, of strong health impairments resulting from the research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2018-03-28 (Estimated); Study Completion 2018-03-28 (Estimated)

PRIMARY OUTCOMES:
Intra ocular measurements differences | 3 years
  Raising intra-abdominal pressure may cause a rise in intraocular pressure. The aim of this research is to examine the changes in IOP before and after the virtual colonoscopy, with the aim to improve the understanding of the relationship between intra-abdominal pressure and IOP.

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual participant data